CLINICAL TRIAL: NCT03762759
Title: Advanced PET-CT Directed Post-Prostatectomy Radiotherapy to Enhance Prostate Cancer Outcomes
Brief Title: Fluciclovine F18 or Ga68-PSMA PET/CT to Enhance Prostate Cancer Outcomes
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Emory University (Other)
Collaborators: Telix Pharmaceuticals (Innovations) Pty Limited (Industry); National Cancer Institute (NCI) (NIH); National Institutes of Health (NIH) (NIH)
Responsible Party: Principal Investigator, Ashesh B Jani, Principal Investigator, Emory University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IRB00106863; NCI-2018-02702 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); RAD4516-18 (Other: Emory University Hospital/Winship Cancer Institute); R01CA226992 (NIH); P30CA138292 (NIH)
Record Dates: First submitted 2018-11-27; First posted 2018-12-04 (Actual); Last update posted 2024-05-17 (Actual); Status verified 2024-05

CONDITIONS: Prostate Adenocarcinoma
MeSH Terms: interventions — fluciclovine F-18; gallium 68 PSMA-11; 68Ga-DKFZ-PSMA-11; Magnetic Resonance Spectroscopy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Arm I (fluciclovine F18, PET/CT) (Experimental): Patients receive fluciclovine F18 IV and undergo positron emission tomography (PET)/computed tomography (CT) over 30 minutes.
  Interventions: Procedure: Computed Tomography; Drug: Fluciclovine F18; Procedure: Positron Emission Tomography
- Arm II (68Ga-PSMA, PET/CT) (Active Comparator): Patients receive gallium Ga68-labeled PSMA-11 IV, wait 60 minutes, then undergo positron emission tomography (PET)/computed tomography (CT) over 30 minutes.
  Interventions: Procedure: Computed Tomography; Radiation: Gallium Ga68-labeled PSMA-11; Procedure: Positron Emission Tomography

INTERVENTIONS:
Procedure: Computed Tomography — Undergo PET/CT
  Other Names: CT; CT scan; Computerized axial tomography; CAT; CAT scan
Drug: Fluciclovine F18 — Given IV
  Other Names: anti-3-[18F]FACBC; Anti-1-Amino-3-[18F]Fluorocyclobutane-1-Carboxylic Acid; FACBC; [18F]FACBC; Axumin
  Arms: Arm I (fluciclovine F18, PET/CT)
Radiation: Gallium Ga68-labeled PSMA-11 — Given IV
  Other Names: 68Ga-PSMA; 68Ga PSMA; [68Ga] Prostate-specific Membrane Antigen 11; 68Ga-DKFZ-PSMA-11; 68Ga-PSMA-HBED-CC
  Arms: Arm II (68Ga-PSMA, PET/CT)
Procedure: Positron Emission Tomography — Undergo PET/CT
  Other Names: PET; PET scan; Proton magnetic resonance spectroscopic imaging

SUMMARY:
This phase II trial studies how well a positron emission tomography (PET)/computed tomography (CT) scan using fluciclovine F18 compared with a PET/CT scan with 68Ga-PSMA works in planning radiation treatments and enhancing outcomes in patients with prostate adenocarcinoma. Fluciclovine F18 and 68Ga-PSMA are types of tracers, called radiotracers, that are injected and can accumulate in tumor cells to develop images of them during a PET/CT scan. It is not yet known whether giving fluciclovine F18 or 68Ga-PSMA may work better in planning radiation treatments and enhancing outcomes in patients with prostate adenocarcinoma.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES

I. Improve the outcomes of post-prostatectomy radiotherapy prostate cancer patients via selection and treatment optimization with advanced molecular imaging with dose escalation.

II. Establish the role of advanced molecular imaging with fluciclovine F18 (fluciclovine [18F]) and gallium Ga68-labeled prostate specific membrane antigen PSMA-11 (68Ga-PSMA) PET/CT in influencing post-prostatectomy radiotherapy decision-making.

III. Establish the role of advanced molecular imaging with fluciclovine 18F or 68Ga-PSMA in altering radiotherapy treatment volumes.

OUTLINE: Patients are randomized to 1 of 2 arms.

ARM I: Patients receive fluciclovine F18 intravenously (IV) and undergo a PET/CT over approximately 30 minutes.

ARM II: Patients receive 68Ga-PSMA IV, wait 60 minutes, then undergo a PET/CT over approximately 30 minutes.

After completion of study treatment, patients are followed up every 6 months for up to 5 years.

ELIGIBILITY:
Inclusion Criteria:

* Adenocarcinoma of the prostate, post radical-prostatectomy
* Detectable prostate-specific antigen (PSA)
* Eastern Cooperative Oncology Group (ECOG)/Zubrod performance status of 0-2
* No definitive findings for skeletal metastasis on technetium 99-m methyl diphosphonate (MDP) or F-18 PET bone scan
* No definitive findings of systemic (extrapelvic) metastasis on CT and/or magnetic resonance (MR) scan of abdomen and pelvis
* Willingness to undergo pelvic radiotherapy

Exclusion Criteria:

* Contraindications to radiotherapy (including active inflammatory bowel disease or prior pelvic radiotherapy)
* Inability to undergo fluciclovine or Ga-PSMA PET-CT
* Definitive findings of systemic metastasis on conventional imaging or biopsy
* Prior invasive malignancy (except non-melanomatous skin cancer) unless disease free for a minimum of 3 years
* Severe acute co-morbidity, defined as follows:

  * Unstable angina and/or congestive heart failure requiring hospitalization in the last 3 months
  * Transmural myocardial infarction within the last 6 months
  * Acute bacterial or fungal infection requiring intravenous antibiotics at the time of registration
  * Chronic Obstructive Pulmonary Disease exacerbation or other respiratory illness requiring hospitalization or precluding study therapy at the time of registration
  * Acquired immune deficiency syndrome (AIDS) based upon current Center for Disease Control (CDC) definition; note, however, that human immunodeficiency virus (HIV) testing is not required for entry into this protocol. The need to exclude patients with AIDS from this protocol is necessary because the treatments involved in this protocol may be significantly immunosuppressive. Protocol-specific requirements may also exclude immunocompromised patients

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 140 (Actual)
Dates: Start 2019-05-10 (Actual); Primary Completion 2025-05-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Disease-free survival | Up to 2 years after study start
  A survival analysis will be conducted on disease-free survival (DFS). The survivor functions for DFS will be estimated with Kaplan and Meier method and plotted. The logrank test will be used to test the difference in DFS of (a) both arms in aggregate with the survivor function on our prior R01 trial and (b) between the two study arms.

SECONDARY OUTCOMES:
Decision to offer radiotherapy | Up to 5 years after study start
  Decision to offer radiotherapy or not between the initial (pre-fluciclovine F18 or 68Ga-PSMA) and final (post-fluciclovine F18 or 68Ga-PSMA) treatment decisions will be compared using the Clopper-Pearson (exact) binomial test.
Decision to treat pelvic nodes | Up to 5 years after study start
  Decision to provide treatment on pelvic nodes or not between the initial (pre-fluciclovine F18 or 68Ga-PSMA) and final (post-fluciclovine F18 or 68Ga-PSMA) treatment decisions will be compared using the Clopper-Pearson (exact) binomial test.
Decision to boost between the initial and final treatment decisions | Up to 5 years after study start
  Decision to boost or not between the initial (pre-fluciclovine F18 or 68Ga-PSMA) and final (post-fluciclovine F18 or 68Ga-PSMA) treatment decisions will be compared using the Clopper-Pearson (exact) binomial test.
Prostate bed clinical target volume (CTV) and planning target volume (PTV) | Up to 5 years after study start
  Paired t-test will be used to compare the target volumes (CTV and PTV) and the planned dose delivered to surrounding bladder, rectum, and penile bulb between the initial (pre-positron emission tomography [PET]) and final (post-PET) radiation treatment plans.
PTV of the rectum (V65, V40) | Up to 5 years after study start
  Spearman's correlation coefficient will be used to measure the correlations of the bladder and rectum dosimetric endpoints (V65, V40) with the grades (0, 1, 2, or 3) of acute genitourinary (GU) or gastrointestinal (GI) toxicity. A Wald test will be used to test the significance level of their correlations. A Cox model will be employed to assess the relationship between the time to late GU or GI toxicity (grade ≥ 2) and the bladder and rectum dosimetric endpoints (V65, V40), respectively.
PTV of the bladder (V65, V40) | Up to 5 years after study start
  Spearman's correlation coefficient will be used to measure the correlations of the bladder and rectum dosimetric endpoints (V65, V40) with the grades (0, 1, 2, or 3) of acute GU or GI toxicity. A Wald test will be used to test the significance level of their correlations. A Cox model will be employed to assess the relationship between the time to late GU or GI toxicity (grade ≥ 2) and the bladder and rectum dosimetric endpoints (V65, V40), respectively.

CONTACTS AND LOCATIONS:
Overall Officials: Ashesh Jani, MD, MSEE, Principal Investigator — Emory University
Locations (3):
- United States (3):
  - Grady Health System, Atlanta, Georgia
  - Emory University Hospital/Winship Cancer Institute, Atlanta, Georgia
  - Emory Saint Joseph's Hospital, Atlanta, Georgia

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Informed Consent Form (2022-10-17): https://cdn.clinicaltrials.gov/large-docs/59/NCT03762759/ICF_000.pdf